CLINICAL TRIAL: NCT01137188
Title: Effect of Weight Loss on Skin Manifestations, Inflammatory Markers and Risk Factor for Comorbidity in Obese Patients With Psoriasis - a Randomized Cross-over Study
Brief Title: Effect of Weight Loss on Psoriasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Peter Jensen, MD, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: H-2-2010-001
Record Dates: First submitted 2010-03-18; First posted 2010-06-04 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-04

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Intensive weight loss program and regular group sessions with clinical dietician. Complete dietary substitution with a low calorie diet containing 800-1000 kcal/day for 8 weeks
  Interventions: Dietary Supplement: Low calorie diet
- No intervention (No Intervention): Study subjects will receive routine dietary counseling for 8 weeks and will cross over to intervention upon completion

INTERVENTIONS:
Dietary Supplement: Low calorie diet — Low calorie diet containing 800-1000 kcal/day
  Arms: Intervention group

SUMMARY:
Controlled data show that obesity is a risk factor for psoriasis and that psoriasis severity is correlated with the degree of overweight. No controlled interventional studies reporting on the effect of weight loss on psoriatic skin manifestations have been published and data from case reports are conflicting.

Patients with psoriasis demonstrate an increased susceptibility to atherosclerotic comorbidities such as arterial hypertension, coronary vascular disease, stroke, hyperlipidemia and type II diabetes and in severe psoriasis there is an increased risk of early death. Lately the role of inflammation in the atherosclerotic process has been highlighted and the link between psoriasis and atherosclerosis may be explained by the concomitant systemic inflammation in psoriasis. Similarly a state of low level inflammation is seen in obesity where macrophages and adipocytes begin to show overlap in function and gene expression. This leads to an increased migration of macrophages into the adipose tissue and an increased secretion of pro-inflammatory cytokines. In summary, these data and theoretical considerations suggest that weight loss in obese patients with psoriasis may improve skin manifestations and reduce the risk of atherosclerotic comorbidity.

ELIGIBILITY:
Inclusion Criteria:

* moderate/severe psoriasis at inclusion or previous to systemic immunosuppressive therapy
* BMI > 27

Exclusion Criteria:

* pregnancy/breast feeding
* diabetes requiring insulin treatment
* severe heart/kidney/liver disease
* gout
* high potassium intake
* obesity due to medical conditions/medications
* use of medical treatment for obesity
* previous bariatric surgery
* intentional/unintentional weight loss up to 3 months prior to inclusion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
PASI | Baseline
  Psoriasis area and severity index
PASI | 4 weeks
  Psoriasis area severity index
PASI | 8 weeks
  Psoriasis area severity index
PASI | 12 weeks
  Psoriasis area severity index
PASI | 16 weeks
  Psoriasis area severity index

SECONDARY OUTCOMES:
Risk factors for comorbidity | Baseline
  Risk factors for comorbidity
Risk factors for comorbidity | 4 weeks
  Risk factors for comorbidity
Risk factors for comorbidity | 8 weeks
  Risk factors for comorbidity
Risk factors for comorbidity | 12 weeks
  Risk factors for comorbidity
Risk factors for comorbidity | 16 weeks
  Risk factors for comorbidity

CONTACTS AND LOCATIONS:
Overall Officials: Lone Skov, MD, phd, Principal Investigator — Copenhagen University Hospital Gentofte, Department of Dermato-venerology
Locations (1):
- Copenhagen University Hospital Gentofte, Department of Dermato-venerology, Hellerup, Denmark

REFERENCES:
- [Derived] Jensen P, Christensen R, Zachariae C, Geiker NR, Schaadt BK, Stender S, Hansen PR, Astrup A, Skov L. Long-term effects of weight reduction on the severity of psoriasis in a cohort derived from a randomized trial: a prospective observational follow-up study. Am J Clin Nutr. 2016 Aug;104(2):259-65. doi: 10.3945/ajcn.115.125849. Epub 2016 Jun 22. PMID 27334236
- [Derived] Jensen P, Zachariae C, Christensen R, Geiker NR, Schaadt BK, Stender S, Astrup A, Hansen PR, Skov L. Effect of weight loss on the cardiovascular risk profile of obese patients with psoriasis. Acta Derm Venereol. 2014 Nov;94(6):691-4. doi: 10.2340/00015555-1824. PMID 24556829
- [Derived] Jensen P, Zachariae C, Christensen R, Geiker NR, Schaadt BK, Stender S, Hansen PR, Astrup A, Skov L. Effect of weight loss on the severity of psoriasis: a randomized clinical study. JAMA Dermatol. 2013 Jul;149(7):795-801. doi: 10.1001/jamadermatol.2013.722. PMID 23752669